CLINICAL TRIAL: NCT06868511
Title: Neuronavigation-assisted Stereotactic Minimally Invasive Puncture Combined With Tenecteplase for the Treatment of Acute Spontaneous Deep Intracerebral Hemorrhage(NAS-TNK)： a Randomized, Outcome-blinded, Multi-center Trial
Brief Title: Neuronavigation-assisted Stereotactic Puncture With Tenecteplase for Acute Intracerebral Hemorrhage
Acronym: NAS-TNK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Dr. Yong Cao, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAS-TNK-ICH
Record Dates: First submitted 2025-03-04; First posted 2025-03-11 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Deep Intracerebral Hemorrhage (ICH)
Keywords: Tenecteplase; Neuronavigation-assisted Stereotactic; Deep intracerebral hemorrhage
MeSH Terms: interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard medical treatment group (Sham Comparator): The standard medical treatment for this group of patients will be provided according to the optimal care standards outlined by the American Heart Association (AHA) for the management of intracerebral hemorrhage.
  Interventions: Drug: Standard medical treatment
- NAS-TNK group (Experimental): This intervention involves neuronavigation-assisted stereotactic (NAS) minimally invasive puncture combined with tenecteplase (TNK). NAS minimally invasive puncture enhances catheter placement precision, reducing complications and improving hematoma evacuation and neurological outcomes. TNK, a third-generation thrombolytic, offers advantages over alteplase (rt-PA) , including a longer half-life for rapid bolus administration and effective thrombolytic effects to dissolve clots and promote hematoma clearance.
  Interventions: Procedure: Neuronavigation-assisted Stereotactic Minimally Invasive Puncture Combined with Tenecteplase

INTERVENTIONS:
Procedure: Neuronavigation-assisted Stereotactic Minimally Invasive Puncture Combined with Tenecteplase — Neuronavigation-assisted stereotactic minimally invasive puncture will enhances catheter placement precision, reducing complications and improving hematoma evacuation and neurological outcomes. TNK, a third-generation thrombolytic will offers advantages over alteplase (rt-PA), including a longer half-life for rapid bolus administration and effective thrombolytic effects to dissolve clots and promote hematoma clearance.
  Arms: NAS-TNK group
Drug: Standard medical treatment — The standard medical treatment for this group of patients will be provided according to the optimal care standards defined by the American Heart Association (AHA) guidelines for intracerebral hemorrhage management
  Arms: Standard medical treatment group

SUMMARY:
Background Minimally invasive puncture surgery followed by thrombolysis has been proven to be an effective approach for managing hypertensive intracerebral hemorrhage. Nevertheless, its impact on improving neurological outcomes remains controversial. The integration of neuronavigation-assisted stereotactic (NAS) technology will significantly help enhance the accuracy of catheter placement, while tenecteplase (TNK), a third-generation thrombolytic agent, with greater potency in lysing platelet-rich clots and heightened specificity for fibrin may improve thrombolysis efficiency. However, the efficacy and safety of combining NAS minimally invasive puncture combined with TNK in reducing disability and mortality rates among patients with acute spontaneous deep intracerebral hemorrhage remain unknown.

Aim To evaluate the efficacy and safety of neuronavigation-assisted stereotactic MIPS combined with TNK thrombolysis （NAS-TNK）in reducing disability and mortality in patients with deep hypertensive intracerebral hemorrhage.

Design NAS-TNK is a randomized, open-label, outcome-blinded multicenter trial, involving 732 participants with acute basal ganglia or thalamic hemorrhage with a hematoma volume ranging from 20-50 mL. This study will evaluate the efficacy and safety of NAS minimally invasive puncture combined with TNK, administered every 24 hours at a dose of 0.009 mg per milliliter of hematoma volume, compared to participants receiving standard medical care. All patients will be followed up for 180 days.

Study outcomes The primary efficacy outcome is the proportion of subjects in the NAS-TNK group with a modified Rankin Scale (mRS) score between 0 and 3 at 180 days. The primary safety outcome is the all-cause death at 30-day.

The NAS-TNK study will help improve our understanding of the benefits of NAS minimally invasive puncture combined with TNK in patients with acute spontaneous deep intracerebral hemorrhage. This ongoing research will provide Level I evidence to guide clinicians in managing acute intracerebral hemorrhage treatment options.

DETAILED DESCRIPTION:
Every year, more than 5 million cases of brain hemorrhage are reported worldwide. Minimally invasive surgery (MIS) has been established as an effective approach for treating acute spontaneous intracerebral hemorrhage and has received endorsement from both international and national clinical guidelines. Randomized controlled trials, such as MISTIE II, MISTIE III, and ENRICH, have demonstrated that procedures involving minimally invasive puncture or endoscopic hematoma evacuation significantly lower mortality rates among patients suffering from intracerebral hemorrhage. Data from these studies indicate that the mortality rate in the minimally invasive treatment groups has decreased from 18% to 26% down to approximately 9% to 19%. Additionally, the 2022 guidelines published by the American Heart Association and the American Stroke Association recommend these minimally invasive techniques as the preferred surgical intervention for patients with hematoma volumes exceeding 20 to 30 milliliters.

Minimally invasive puncture surgery (MIPS) combined with thrombolysis is particularly favored for its simplicity and broad applicability. This technique effectively aids in the evacuation of hematomas and alleviates pressure in cases of deep acute spontaneous intracerebral hemorrhages, all while minimizing the risk of iatrogenic injury and maximizing the protection of neural tissue. Although MIPS has shown promising outcomes in reducing procedure-related trauma, the long-term effectiveness of this method in preventing neurological deficits remains a subject of ongoing debate. Recent findings from the MISTIE III trial shed light on this issue. In this trial, the MISTIE group exhibited a mortality rate of 15% at 180 days, a significant reduction compared to the 23% observed in the standard care group (p=0.033). Furthermore, at 365 days, 45% of patients treated with MIPS achieved a modified Rankin Scale (mRS) score of 0 to 3, indicating favorable functional outcomes, compared to 41% in the standard medical care group, with no statistically significant difference observed between the two groups.

Nonetheless, subgroup analyses from the MISTIE III trial indicated that patients who underwent surgical intervention and achieved a hematoma reduction to less than 15 mL experienced significantly improved functional outcomes compared to those who received conservative treatment. This suggests that, in clinically stable patients, more aggressive and rapid removal of intracerebral hematomas may effectively lower the risk of mortality and enhance functional outcomes. Therefore, conducting trials that focus on rapid and extensive removal of hematoma volumes combined with MIPS would be beneficial in achieving better functional results.

The precise placement of the catheter tip within the hematoma is critical for the efficient and rapid evacuation of intracerebral hematoma. The thrombolytic agent delivered from the catheter tip relies on gravity to infiltrate and interact with the clot, thereby facilitating its dissolution. Simultaneously, the liquefied hematoma fluid is drained through the catheter tip. Neuronavigation-assisted stereotactic (NAS) technology can significantly enhance the accuracy of catheter tip placement, thereby reducing the risk of iatrogenic injuries and complications.

Tenecteplase (TNK), a third-generation thrombolytic agent derived from alteplase (rt-PA), offers several advantages over its predecessor. Its extended half-life allows for rapid administration via bolus infusion, providing logistical benefits compared to rt-PA. Additionally, TNK demonstrates increased resistance to inactivation by plasminogen activator inhibitor-1, resulting in a greater potency for lysing platelet-rich clots. Its heightened specificity for fibrin may also contribute to a reduction in hemorrhagic complications, especially those associated with systemic bleeding. These benefits have been evidenced in studies focused on conditions such as myocardial infarction and acute ischemic stroke. TNK has also shown effective thrombolytic effects, aiding in the dissolution of clots and promoting hematoma clearance. However, the efficacy and safety of combining NAS-assisted minimally invasive puncture with TNK (NAS-TNK) to reduce disability and mortality rates in patients with acute spontaneous deep intracerebral hemorrhage remain uncertain.

The NAS-TNK trial is designed to explore the impact of precise, rapid, and efficient clearance of hematoma volumes on the improvement of neurological function in patients. This multicenter, randomized, outcome-blinded study will evaluate the efficacy and safety of neuronavigation-assisted stereotactic MIPS combined with TNK thrombolysis in reducing disability and mortality rates in patients suffering from deep hypertensive intracerebral hemorrhage. This paper presents the design of the NAS-TNK trial and outlines its protocol in detail.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and <80 years.
2. Symptoms must have manifested within 24 hours prior to the diagnostic CT (dCT) scan. Cases with an indeterminate onset time are excluded. For patients who present symptoms upon sleeping, the last known time they were well should be used.
3. Acute spontaneous deep intracerebral hemorrhage (ICH) occurring in the basal ganglia or thalamus, with a volume between 20-50 mL as measured by ABC/2 method with radiographic imaging (CT, etc.).
4. Glasgow Coma Scale (GCS) score of 5-14.
5. Stability CT scan done at least 6 hours after diagnostic CT showing clot stability (growth<5 mL as measured by ABC/2 method).
6. Randomization should occur within 6 to 24 hours after the diagnostic CT.
7. Systolic blood pressure (SBP) less than 180 mmHg maintained for a duration of six hours, documented proximate to the randomization time point.
8. Historical Rankin score of 0 or 1.

Exclusion Criteria:

1. Lobar or subtentorial hemorrhage, including posterior fossa hemorrhage and cerebellar hemorrhage.
2. Stability CT scan done at least 6 hours after diagnostic CT showing clot instability (growth ≥5 mL as measured by ABC/2 method).
3. Intraventricular hemorrhage necessitating intervention to address mass effect or midline shift attributable to trapped ventricle syndrome secondary to intraventricular hemorrhage (IVH)-related casting.
4. Hemorrhage attributable to other cerebrovascular pathologies, including but not limited to ruptured aneurysm, arteriovenous malformation (AVM), vascular anomalies, moyamoya disease, hemorrhagic transformation of an ischemic infarct, or recurrence of a recent hemorrhage within the past year, as diagnosed through radiographic imaging.
5. Patients presenting with an unstable intracranial mass or progressive intracranial compartment syndrome.
6. Thalamic hemorrhages exhibiting evident extension into the midbrain, accompanied by oculomotor nerve palsy or pupils that are dilated and non-reactive. Other supranuclear gaze abnormalities do not constitute exclusion criteria.
7. Irreversible impairment of brainstem function, characterized by bilateral fixed and dilated pupils, extensor motor posturing, and a Glasgow Coma Scale (GCS) score of ≤ 4.
8. Indications for craniotomy in patients include: 1) progressive impairment of consciousness; 2) presence of brain herniation, with signs related to cerebellar tonsil herniation or temporal lobe gyrus herniation; 3) hematoma located within 1 cm of the cortical surface.
9. CT evidence suggesting a high risk of rebleeding, such as spot sign.
10. Platelet count <100,000/mL; INR >1.4.
11. Any irreversible coagulation disorders (e.g., hemophilia, von Willebrand disease, use of anticoagulants such as warfarin) or known clotting disorders (e.g., hypercoagulable states).
12. Inability to maintain INR ≤1.4 using short-acting and long-acting procoagulants (e.g., recombinant human coagulation factor VIIa, fresh frozen plasma, vitamin K, etc.).
13. Subjects necessitating long-term anticoagulation therapy are excluded from participation. Reversal of anticoagulation is permissible for medically stable patients who can feasibly tolerate the short-term risks associated with reversal. Patients must not require Coumadin (warfarin) or other anticoagulants during the initial 30-day period.
14. Prior to the onset of symptoms, anticoagulants such as dabigatran, apixaban, or rivaroxaban, as well as treatments like tirofiban, ticagrelor, cilostazol, or clopidogrel, were used.
15. Internal bleeding involving the retroperitoneal, gastrointestinal, or genitourinary system, or respiratory tract bleeding.
16. Superficial or surface bleeding, observed mainly at vascular puncture and access sites (e.g., venous cutdowns, arterial punctures, etc.) or site of recent surgical intervention.
17. Positive urine or serum pregnancy test in pre-menopausal female subjects without a documented history of surgical sterilization.
18. Allergy/sensitivity to TNK.
19. Prior enrollment in the study.
20. Engagement in a concurrent interventional clinical investigation or trial. Patients enrolled in observational, natural history, or epidemiological studies that do not involve any form of intervention remain eligible.
21. Not expected to survive until the day 180 visit due to co-morbidities, or having DNR/DNI status (Do-Not-Resuscitate and Do-Not-Intubate) prior to randomization.
22. The presence of any concurrent serious illness that could confound outcome assessments, including but not limited to hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, or hematologic disorders.
23. Patients with mechanical heart valves are excluded. The presence of bioprosthetic valve(s) is permissible.
24. Known risk for embolization, including history of left heart thrombus, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. Atrial fibrillation without mitral stenosis is permitted.
25. Any other condition that, in the investigator's judgment, would present a significant risk to the subject if the investigational therapy were to be initiated.
26. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
27. Patients deemed by the investigator to have unstable conditions that may benefit from other treatments.
28. Patients requesting conservative treatment or standard craniotomy microsurgery treatment.
29. The subject or their legal guardian/representative demonstrates an inability or lack of willingness to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 732 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) score of 0-3 at 180 days. | 180 ±14 days
  The primary efficacy outcome is the proportion of patients achieving a favorable functional outcome, defined as a modified Rankin Scale (mRS) score of 0-3 at 180 days.

SECONDARY OUTCOMES:
Dichotomized eGOS (extended Glasgow Outcome Scale) score at 180 days: 4-8 (good) vs. 1-3(poor) | 180 ± 14 days
  Dichotomized eGOS (extended Glasgow Outcome Scale) score at 180 days: 4-8 (good) vs. 1-3 (poor). The eGOS is scored as: 1=Death, 2=Vegetative state, 3=Lower severe disability, 4=Upper severe disability, 5=Lower moderate disability, 6=Upper moderate disability, 7=Lower good recovery, 8=Upper good recovery.
All-cause death at 180 days | 180 ± 14 days
  All-cause death at 180 days
Dichotomized, modified Rankin Scale (mRS) Score 0-3 vs. 4-6 at 90 days. | 90 ± 7 days
  Proportion of patients with mRS of 0-3 (good functional status) at 90 days. The mRS is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death. Dichotomized scores are: 0-3=No symptoms to moderate disability requiring some assistance; 4-6=Moderately severe disability requiring complete assistance to death.
Dichotomized graded modified Rankin Scale (mRS) score at 180 days : 0-2 vs. 3-6. | 180 ± 14 days
  Dichotomized graded modified Rankin Scale (mRS) score at 180 days post-hemorrhage: 0-2 vs. 3-6. The mRS is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death. Dichotomized scores are: 0-2=No symptoms to slight disability; 3-6=Moderate disability requiring some assistance to death.
Ordinal graded modified Rankin Scale (mRS) score (0-6) at 180 days. | 180 ± 14 days
  Ordinal graded modified Rankin Scale (mRS) score (0-6) at 180 days. The mRS is scored from: 0=No symptoms at all, 1=No significant disability, 2=Slight disability, 3=Moderate disability, 4=Moderately severe disability, 5=Severe disability and 6=death.
Barthel Index (BI) assessment at 180 days. | 180 ±14 days.
  Barthel Index assessment at 180 days. The Barthel Index (BI) assesses ten functional tasks of daily living, and each task provides a measure for level of independence. Scores range from 0 and 100, with a higher score indicating greater independence.
Extended Glasgow Outcome (eGOS) assessment at 180 days. | 180 ± 14 days
  Extended Glasgow Outcome (eGOS) assessment at 180 days. The extended Glasgow Outcome Scale (eGOS) is a global scale for functional outcome with eight categories: 1 - Death, 2 - Vegetative State, 3 - Lower Severe Disability, 4 - Upper Severe Disability, 5 - Lower Moderate Disability, 6 - Upper Moderate Disability, 7 - Lower Good Recovery, 8 - Upper Good Recovery.
The change of the National Institutes of Health Stroke Scale (NIHSS) at 5-7 days or discharge if earlier from baseline. | 5-7 days
  The change of the National Institutes of Health Stroke Scale (NIHSS) at 5-7 days or discharge if earlier from baseline. Patients with a NIHSS score of less than 6 are considered to have a good recovery. The NIHSS is a 11-item scale that assesses language, motor function, sensory loss, consciousness, visual fields, extraocular movements, coordination, neglect, and speech. It is scored from 0 (no stroke symptoms) to 42 (severe stroke).
Safety/Mortality - All-cause death at 30 days | Within 30 days.
  All-cause death at 30 days
Safety/Mortality - All-cause death at 7 days | Within 7 days
  All-cause death at 7 days
Safety/Mortality - Symptomatic rebleeding within 6 days | Within 6 days
  Symptomatic rebleeding events within 6 days post-randomization (defined as a persistent decrease in GCS motor score by more than 2 points, with a CT scan showing a new hematoma with a CT value greater than 72 HU and a volume exceeding 5 ml within the hematoma cavity and surrounding area compared to the prior scan).
Safety/Mortality - Intracranial bacterial infection within 30 days | Within 30 days
  Intracranial bacterial infection within 30 days.
Safety/Mortality - Total Adverse Events (AEs) within 30 and 180 days | Within 30 and 180 days
  Total Adverse Events (AEs) across all coded organ systems that occurred within 30 and 180 days.
Safety/Mortality - Total Serious Adverse Events (SAEs) within 30 and 180 days | Within 30 and 180 days
  Total Serious Adverse Events (SAEs) within 30 and 180 days.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cao, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: Undecided